CLINICAL TRIAL: NCT06901531
Title: A Phase 3, Double-blind, Randomized Study of Zolbetuximab in Combination With Pembrolizumab and Chemotherapy (CAPOX or mFOLFOX6) in First-line Treatment of Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma in Participants Whose Tumors Are HER2-negative, Claudin (CLDN) 18.2-positive and Programmed Death-ligand 1 (PD-L1)-Positive
Brief Title: A Study of Zolbetuximab Together With Pembrolizumab and Chemotherapy in Adults With Gastric Cancer
Acronym: LUCERNA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8951-CL-0305; 2024-519773-19 (Registry Identifier: CTIS (EU)); jRCT2031250021 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); CTR20253090 (Registry Identifier: ChinaDrugTrials.org.cn)
Expanded Access: NCT06048081 (Available)
Record Dates: First submitted 2025-03-27; First posted 2025-03-30 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Unresectable Gastroesophageal Junction (GEJ) Adenocarcinoma or Cancer; Locally Advanced Unresectable Gastric Adenocarcinoma or Cancer; Metastatic Gastric Adenocarcinoma or Cancer; Metastatic Gastroesophageal Junction (GEJ) Adenocarcinoma
Keywords: Locally Advanced Unresectable Gastroesophageal Junction (GEJ) Adenocarcinoma Cancer; Locally Advanced Unresectable Gastric Adenocarcinoma Cancer; Metastatic Gastric Adenocarcinoma Cancer; Metastatic Gastroesophageal Junction (GEJ) Adenocarcinoma; Claudin 18.2; PD-L1; Human epidermal growth factor receptor 2 (HER2) Negative; zolbetuximab
MeSH Terms: conditions — Adenocarcinoma; Neoplasms | interventions — zolbetuximab; pembrolizumab; Capecitabine; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: zolbetuximab in combination with pembrolizumab and chemotherapy (Experimental): Participants will receive zolbetuximab as an intravenous (via a vein) infusion at 800 mg/m2 loading dose at C1D1 followed by subsequent doses of 400 mg/m2 every 2 weeks; or 800 mg/m2 loading dose at C1D1 followed by subsequent doses of 600 mg/m2 every 3 weeks, followed by an intravenous infusion of pembrolizumab at a dose of 200 mg every 3 weeks or 400 mg every 6 weeks. Participants will then receive chemotherapy over 4 or more cycles of either up to 8 CAPOX treatments (oxaliplatin: 130 mg/m2 once every 3 weeks, capecitabine: 1000 mg/m2 twice daily on days 1 through 14 and days 22 through 35 of each cycle), or, up to 12 mFOLFOX6 treatments (oxaliplatin: 85 mg/m2, Folinic acid (leucovorin/local equivalent): 400 mg/m2, 5-FU bolus: 400 mg/m2, 5-FU infusion: 2400 mg/m2) once every 2 weeks (or components of mFOLFOX6 if some components are discontinued due to toxicity). The choice of chemotherapy for each participant is based on investigator's judgment. Each cycle is approximately 42 days.
  Interventions: Drug: zolbetuximab; Drug: Pembrolizumab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Folinic acid (leucovorin or local equivalent); Drug: 5-fluorouracil (5-FU)
- Arm B: Placebo in combination with pembrolizumab and chemotherapy (Active Comparator): Participants will receive matching placebo as an intravenous (via a vein) infusion followed by an intravenous infusion of pembrolizumab at a dose of 200 mg every 3 weeks or 400 mg every 6 weeks. Participants will then receive chemotherapy over 4 or more cycles of either up to 8 CAPOX treatments (oxaliplatin: 130 mg/m2 once every 3 weeks, capecitabine: 1000 mg/m2 twice daily on days 1 through 14 and days 22 through 35 of each cycle), or, up to 12 mFOLFOX6 treatments (oxaliplatin: 85 mg/m2, Folinic acid (leucovorin/local equivalent): 400 mg/m2, 5-FU bolus: 400 mg/m2, 5-FU infusion: 2400 mg/m2) once every 2 weeks (or components of mFOLFOX6 if some components are discontinued due to toxicity). The choice of chemotherapy for each participant is based on investigator's judgment. Each cycle is approximately 42 days.
  Interventions: Drug: Pembrolizumab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Folinic acid (leucovorin or local equivalent); Drug: 5-fluorouracil (5-FU); Drug: Placebo

INTERVENTIONS:
Drug: zolbetuximab — Participants will receive an IV infusion of zolbetuximab on Cycle 1 Day 1 (C1D1) followed by subsequent IV infusion every 2 weeks or every 3 weeks.
  Other Names: IMAB362; VYLOY
  Arms: Arm A: zolbetuximab in combination with pembrolizumab and chemotherapy
Drug: Pembrolizumab — Participants will receive an IV infusion of pembrolizumab every 3 weeks or every 6 weeks.
Drug: Capecitabine — Participants receiving CAPOX regimen of chemotherapy will receive capecitabine Tablet twice daily orally on days 1 through 14 and days 22 through 35 of each cycle.
Drug: Oxaliplatin — Participants receiving CAPOX or mFOLFOX6 regimen of chemotherapy will receive an IV infusion of oxaliplatin once every 2 or 3 weeks.
Drug: Folinic acid (leucovorin or local equivalent) — Participants receiving mFOLFOX6 regimen of chemotherapy will receive an IV infusion of Folinic acid (leucovorin or local equivalent) once every 2 weeks.
Drug: 5-fluorouracil (5-FU) — Participants receiving mFOLFOX6 regimen of chemotherapy will receive an IV infusion, or IV bolus of 5-FU once every 2 weeks.
Drug: Placebo — Participants will receive an IV infusion of placebo (0.9% of sodium chloride) on C1D1 followed by subsequent IV infusion every 2 weeks or every 3 weeks.
  Arms: Arm B: Placebo in combination with pembrolizumab and chemotherapy

SUMMARY:
Zolbetuximab is being studied in people with cancer in and around the stomach or where the food pipe (esophagus) joins the stomach, called gastroesophageal junction (GEJ) cancer. Zolbetuximab with chemotherapy may be used to treat stomach and GEJ cancer when the cancer cells do not have a protein called HER2 (human epidermal growth factor receptor 2) on their surface (HER2-negative) but do have a protein called Claudin 18.2 (Claudin 18.2-positive). Zolbetuximab is thought to work by attaching to the Claudin 18.2 protein in their tumor, which switches on the body's immune system to attack the tumor. Certain stomach and GEJ cancers may be treated with immunotherapy, which helps the body's immune system fight cancer. This study will give more information about how well zolbetuximab works when given with an immunotherapy medicine called pembrolizumab and chemotherapy. In this study, adults with stomach cancer or GEJ cancer will either be given zolbetuximab with pembrolizumab and chemotherapy or a placebo with pembrolizumab and chemotherapy. A placebo looks like zolbetuximab but doesn't have any medicine in it.

The main aim of the study is to check how long people with stomach cancer and GEJ cancer live after treatment with zolbetuximab with pembrolizumab and chemotherapy compared to placebo with pembrolizumab and chemotherapy.

Adults with locally advanced unresectable or metastatic stomach cancer or GEJ cancer can take part. Locally advanced means the cancer has spread to nearby tissue. Unresectable means the cancer cannot be removed by surgery. Metastatic means the cancer has spread to other parts of the body. A tumor sample (biopsy) of their cancer will have the Claudin 18.2 protein, PD-L1 protein, and be HER2-negative. They may have been previously treated with certain standard therapies. People cannot take part if they need to take medicines to suppress their immune system, have blockages or bleeding in their gut, have specific uncontrollable cancers such as symptomatic or untreated cancers in the nervous system, or have a specific heart condition, or infections.

The study treatments are either zolbetuximab with pembrolizumab and chemotherapy, or placebo with pembrolizumab and chemotherapy. People who take part will receive just 1 of the study treatments by chance. The people in the study and the study doctors will not know who takes which of the study treatments. Study treatment will be given in 6-week (42-day) cycles. The study treatment is mainly given to people slowly through a tube into a vein. This is called an infusion. People will receive study treatment as follows: Zolbetuximab or placebo: 1 infusion every 2 or 3 weeks (2 or 3 infusions in a cycle) together with: Chemotherapy (1 of the following types of chemotherapy): 1. CAPOX (capecitabine and oxaliplatin): 1 infusion of oxaliplatin every 3 weeks (2 infusions in a cycle). People will also take 1 tablet of capecitabine twice a day for 2 weeks (14 days) at the start of each cycle (Day 1) and again in the middle of each cycle (Day 22). After 8 study treatments people will receive capecitabine only. 2. Modified FOLFOX6 or mFOLFOX6 (5-fluorouracil, folinic acid and oxaliplatin): 1 infusion every 2 weeks (3 infusions in a cycle). After 12 study treatments people will receive folinic acid and fluorouracil only, instead of mFOLFOX6. Pembrolizumab: 1 infusion every 3 or 6 weeks (1 or 2 infusions in a cycle). People can be in the study and will receive study treatment until their cancer worsens, they cannot tolerate the study treatment, or they need to start another cancer treatment. People may receive pembrolizumab for up to 2 years. People will visit the clinic on certain days to receive their study treatment and have health checks. The study doctors will check if people had any medical problems from taking zolbetuximab or the other study treatments. On some visits they will have scans to check for any changes in their cancer. People will have the option of giving a tumor sample if they stop treatment because their cancer has worsened. People will visit the clinic after they stop their study treatment. People will be asked about any medical problems and will have a health check. People will continue to have scans every 9 or 12 weeks to check for any changes in their cancer. They will have telephone health checks every 3 months. The number of visits and checks done at each visit will depend on the health of each person and whether they completed their study treatment or not.

DETAILED DESCRIPTION:
Zolbetuximab (Vyloy), has received marketing approval in Japan. The study is considered a post marketing study in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically confirmed gastric or Gastroesophageal Junction (GEJ) adenocarcinoma.
* Participant has radiographically confirmed, locally advanced, unresectable or metastatic disease within 28 days prior to randomization.
* Participant has radiologically evaluable disease (measurable and/or nonmeasurable) according to Response Evaluation Criteria in Solid Tumors (RECIST) V1.1, ≤ 28 days prior to randomization. For participants with only 1 evaluable lesion and prior radiotherapy ≤ 3 months before randomization, the lesion must either be outside the field of prior radiotherapy or have documented progression following radiation therapy.
* Participant has Eastern Cooperative Oncology Group Performance Status (ECOG) performance status 0 to 1.
* Participant has predicted life expectancy ≥ 12 weeks.
* Participant must be a candidate to receive mFOLFOX6 or CAPOX and pembrolizumab.
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of child bearing potential (WOCBP)
  * WOCBP who has a negative urine or serum pregnancy test at screening (Specific to Japan: with a medical interview), and agrees to follow the contraceptive guidance from the time of informed consent through at least 9 months after the final oxaliplatin administration and 6 months after the final administration of all other study intervention.
  * Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 5 half-lives (at least 9 months after the final oxaliplatin administration and 6 months after final study intervention administration).
  * Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period, and for 9 months after the final administration of oxaliplatin and for 6 months after final administration of all other study interventions.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period, and for 6 months after final investigational study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 6 months after the final investigational study intervention administration.
* Male participant must not donate sperm during the treatment period and for 6 months after the final investigational study intervention administration
* Participant has a Human Epidermal Growth Factor Receptor 2 (HER2) -negative tumor.
* Participant's tumor expresses Claudin18.2 (CLDN18.2) in ≥ 75% of tumor cells demonstrating moderate to strong membranous staining as determined by central immunohistochemistry (IHC) testing.
* Participant's tumor expresses Programmed death ligand (PD-L1) combined positive score (CPS) ≥ 1 as determined by central IHC testing.
* Participants with known microsatellite instability-high or mismatch repair deficient status may enroll as long as they meet the PD-L1 positivity criteria.
* Participant must meet all of the criteria based on the centrally or locally analyzed laboratory tests collected within 14 days prior to randomization. In case of multiple central laboratory data within this period, the most recent data should be used.
* Participant agrees not to participate in another interventional study while receiving study intervention in the present study.

Exclusion Criteria:

* Participant has prior severe allergic reaction or intolerance to zolbetuximab or other monoclonal antibodies, pembrolizumab, mFOLFOX6 or CAPOX.
* Participant has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent recurrent vomiting.
* Participant has significant gastric bleeding and/or untreated gastric ulcers that would preclude the participant from participation.
* Participant has unresolved pneumonitis or history of non-infectious pneumonitis such as immune-related pneumonitis, radiation induced pneumonitis.
* Participant has history of central nervous system metastases and/or carcinomatous meningitis from gastric/GEJ cancer.
* Participant has a known history of a positive test for Human Immunodeficiency Virus (HIV) infection or known active Hepatitis B Surface Antigen (positive HBsAg) or hepatitis C infection. NOTE: Screening for these infections should be conducted per local requirements.

  * For participants who are negative for HBsAg, but hepatitis B core antibody (HBcAb) positive, a hepatitis B DNA test will be performed and if positive the participant will be excluded.
  * Participants with positive Hepatitis C virus (HCV) serology, but negative HCV RNA test results are eligible.
  * Participants treated for HCV with undetectable viral load results are eligible.
* Participant has active infection requiring systemic therapy that has not completely resolved within 7 days prior to randomization.
* Participant has active autoimmune disease that has required systemic treatment within the past 3 months prior to randomization.
* Participant has a clinically significant disease or comorbidity that may adversely affect the safe delivery of treatment within this study or make the participant unsuitable for study participation.
* Participant has another malignancy for which treatment is required.
* Participant has known Dihydropyrimidine Dehydrogenase (DPD) deficiency (screening for DPD deficiency should be conducted per local requirements).
* Participant has known peripheral neuropathy > grade 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the participant ineligible).
* Participant has sinusoidal obstruction syndrome, formerly known as veno-occlusive disease, if present, should be stable or improving.
* Participant has significant cardiovascular disease, including any of the following:

  * Congestive heart failure (defined as New York Heart Association Class III or IV), myocardial infarction, unstable angina, coronary angioplasty, coronary stenting, coronary artery bypass graft, cerebrovascular accident or hypertensive crisis within 6 months prior to randomization.
  * History of clinically significant ventricular arrhythmias (i.e., sustained; ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes).
  * QTc interval > 450 msec for male participants; QTc interval > 470 msec for female participants.
  * History or family history of congenital long QT syndrome.
  * Cardiac arrhythmias requiring anti-arrhythmic medications (participants with rate controlled atrial fibrillation for > 1 month prior to randomization are eligible).
* Participant has ongoing or previous interstitial lung disease, active diverticulitis or peptic ulcerative disease, or solid organ or stem cell transplant or other uncontrolled or clinically significant medical disorders.
* Participant has type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy or skin disorders (e.g., vitiligo, psoriasis or alopecia) not requiring systemic treatment are allowed.
* Participant has received prior systemic chemotherapy and/or immunotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma, except for a maximum of 1 treatment course of mFOLFOX6 (day 1 to 14) or CAPOX (day 1 to 21) with or without pembrolizumab. However, participants may have received either neo-adjuvant or adjuvant chemotherapy, immunotherapy or other systemic anticancer therapies as long as it was completed at least 6 months prior to randomization. Participant may have received treatment with herbal medications that have known antitumor activity > 28 days prior to randomization.
* Participant has received systemic immunosuppressive therapy, including systemic corticosteroids 14 days prior to randomization. Participants using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day of prednisone), receiving a single-dose of systemic corticosteroids or receiving systemic corticosteroids as premedication for radiologic imaging contrast use are allowed.
* Participant has had major surgical procedure ≤ 28 days before randomization and has not completely recovered from the surgical procedure ≤ 14 days before randomization.
* Participant has received radiotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma ≤ 14 days prior to randomization and has NOT recovered from any related toxicity. Palliative radiotherapy is allowed and must be completed > 14 days prior to randomization.
* Participant has received prior CLDN18.2 agents.
* Participant received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.
* Participant has received other investigational agents or devices concurrently or within 28 days prior to randomization or within 5 half-lives of the investigational medicinal product (IMP), whichever is longer.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has any concurrent disease, infection, or co-morbid condition that interferes with the ability of the participant to participate in the study, which places the participant at undue risk or complicates the interpretation of data.
* Treatment with brivudine, sorivudine or their chemically related analogues within 28 days prior to randomization or within 5 half-lives of the IMP, whichever is shorter, is strictly prohibited.
* Pernicious anemia or other anemias due to vitamin B12 deficiency.
* Participant has a known history of a positive test for tuberculosis or known active tuberculosis infection. NOTE: Screening for these infections should be conducted per local requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 72 months
  OS is defined as the time from the date of randomization until the date of death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 72 Months
  Defined as the time from the date of randomization until the date of radiologic disease progression [investigator-assessed per Response Evaluation Criteria in Solid Tumors (RECIST) V1.1] or death from any cause, whichever is earlier.
Objective Response Rate (ORR) | Up to 57 Months
  Defined as the proportion of participants who have a Best Overall Response (BOR) or Complete Response (CR) or Partial Response (PR) as investigator assessed per RECIST V1.1.
Duration of Response (DOR) | Up to 72 Months
  Defined as the time from the date of the first response (CR/PR) until the date of disease progression as investigator-assessed per RECIST V1.1 or date of death from any cause, whichever is earlier.
Number of participants with adverse Events (AEs) | Up to 57 Months
  Adverse events (AEs) will coded using MedDRA. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the comparator, if applicable, and events related to the (study) procedures.
Number of participants with electrocardiograms (ECG) abnormalities and/or AEs | Up to 57 Months
  Number of participants with potentially clinically significant ECG values.
Number of Participants with Vital Sign abnormalities and/or AEs | Up to 57 Months
  Number of participants with potentially clinically significant vital sign values.
Number of participants at each grade of Eastern Cooperative Oncology Group (ECOG) performance status score | Up to 57 Months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.
Number of participants with laboratory assessments abnormalities and/ or AEs | Up to 57 Months
  Number of participants with potentially clinically significant laboratory values.
Pharmacokinetics (PK) of zolbetuximab in serum: End of Infusion Concentration | Up to 57 Months
  Concentration will be derived from the PK serum samples collected at time of end of infusion.
Pharmacokinetics (PK) of zolbetuximab in serum: Concentration Immediately Prior to Dosing at multiple dosing (Ctrough) | Up to 57 Months
  Ctrough will be derived from the PK serum samples collected.
Number of participants with positive antidrug antibodies (ADA) to zolbetuximab | Up to 57 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (169):
- United States (20):
  - Yale University School of Medicine, New Haven, Connecticut
  - Franciscan Health Oncology and Hematology Specialists, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Saint Elizabeth Medical Center Edgewood, Edgewood, Kentucky
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Metro Minnesota Community Oncology Research Consortium (MMCORC), Saint Louis Park, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - NYU Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - The University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology-Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - The Center For Cancer And Blood Disorders (Texas Cancer Care), Fort Worth, Texas
  - Houston Methodist Cancer Center, Houston, Texas
- Australia (2):
  - AU61004, Brisbane, Queensland
  - AU61003, Clayton, Victoria
- Belgium (4):
  - BE32002, Bonheiden
  - BE32001, Brussels
  - BE32003, Ghent
  - BE32004, Liège
- China (9):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Sun Yat-sen University - Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital - Oncology, Zhenngzhou, Henan
  - Hubei Cancer Hospital - Oncology, Wuhan, Hubei
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Renji Hospital Shanghai Jiaotong Univ School of Medicine, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Affiliated Hospital of Hebei University, Baoding
- CZ42004, Prague, Czechia
- France (18):
  - FR33016, Bordeaux
  - FR-33008, Brest
  - FR33012, Caen
  - FR33009, Carassonne
  - FR33002, Lille
  - FR33007, Lille
  - FR33014, Lyon
  - FR33017, Lyon
  - FR33020, Montpellier
  - FR33018, Nice
  - FR33003, Paris
  - FR33010, Paris
  - FR33013, Paris
  - FR33015, Plérin
  - FR33004, Poitiers
  - FR33006, Rouen
  - FR33019, Saint Herbian Cedex
  - FR33011, Strasbourg
- Germany (3):
  - DE49002, Saarbrücken
  - DE49011, Schweinfurt
  - DE49016, Wolfsburg
- Italy (14):
  - IT39017, Bologna
  - IT39009, Brescia
  - IT39006, Cermona
  - IT39011, Florence
  - IT39007, Meldola
  - IT-39020, Milan
  - IT39012, Milan
  - IT39018, Milan
  - IT-39015, Pisa
  - IT39004, Reggio Emilia
  - IT39001, Rome
  - IT39003, Torrette Di Ancona
  - IT39022, Udine
  - IT39002, Verona
- Japan (22):
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kyushu University Hospital (Hematology, Oncology & Cardiovascular medicine), Fukuoka, Fukuoka
  - Kyushu University Hospital(Gastrointestinal Surgery), Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi-shi, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kagawa University Hospital, Kida-gun, Kagawa-ken
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Kanagawa Cancer Ctr Hospital, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Saitama Cancer Center, Kitaadachi-gun Ina-machi, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- Lithuania (2):
  - LT37001, Kaunas
  - LT37002, Vilnius
- Netherlands (2):
  - NL-31002, Leeuwarden
  - NL31001, Nijmegen
- Poland (6):
  - PL48005, Lubin, Lubusz Voivodeship
  - PL48004, Warsaw, Masovian Voivodeship
  - PL48001, Brzozów, Woj Podkarpackie
  - PL48008, Olsztyn
  - PL48002, Przemyśl
  - PL48007, Warsaw
- Portugal (3):
  - PT35106, Almada
  - PT35103, Braga
  - PT35104, Guimarães
- Romania (8):
  - RO40008, Bucharest
  - RO40001, Cluj-Napoca
  - RO40005, Cluj-Napoca
  - RO40006, Cluj-Napoca
  - RO40003, Craiova
  - RO40002, Floreşti
  - RO40007, Iași
  - RO40004, Timișoara
- South Korea (15):
  - KR82011, Goyang-si, Gyeonggi-do
  - KR82007, Seongnam-si, Gyeonggi-do
  - KR82013, Suwon, Gyeonggi-do
  - KR82015, Suwon, Gyeonggi-do
  - KR82014, Hwasungun, Joellanamdo
  - KR82009, Cheongju-si, North Chungcheong
  - KR82003, Seocho-gu, Seoul
  - KR82004, Daegu
  - KR82005, Incheon
  - KR82001, Seoul
  - KR82002, Seoul
  - KR82006, Seoul
  - KR82008, Seoul
  - KR82010, Seoul
  - KR82012, Seoul
- Spain (25):
  - ES34022, Elche, Alicante
  - ES34023, San Cugat Del Valles Barcelona, Cataluyna
  - ES34019, Madrid, Madrid
  - ES34027, Madrid, Madrid
  - ES34002, Navarra, Pamplona
  - ES34005, A Coruña
  - ES34006, Barcelona
  - ES34009, Barcelona
  - ES34010, Barcelona
  - ES34011, Barcelona
  - ES34024, Barcelona
  - ES34026, Barcelona
  - ES34021, El Palmar
  - ES34014, Lleida
  - ES34003, Madrid
  - ES34008, Madrid
  - ES34016, Madrid
  - ES34017, Madrid
  - ES34030, Murcia
  - ES34013, Pozuelo de Alarcón
  - ES34029, Santiago de Compostela
  - ES34012, Seville
  - ES34025, Seville
  - ES34004, Valencia
  - ES34007, Valencia
- Taiwan (4):
  - TW-88603, Dawan, Taiwan
  - TW88604, Kaohsiung City
  - TW88601, Taichung
  - TW88606, Tainan
- United Kingdom (11):
  - GB44010, Cottingham, East Riding Of Yorkshire
  - UK44001, Bristol
  - GB44002, Coventry
  - UK44006, Dundee
  - GB44004, Glasgow
  - GB-44005, London
  - UK44011, London
  - UK44014, London
  - UK44015, London
  - UK44016, London
  - UK44009, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as compounds terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/